CLINICAL TRIAL: NCT00425009
Title: Effects of Berberine on Improvement of Glucose and Lipid Metabolism in Patients With Type 2 Diabetes
Brief Title: Therapeutic Effects of Berberine in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-2002-Clin4
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2007-01-22 (Estimated); Status verified 2007-01

CONDITIONS: Type 2 Diabetes
Keywords: Berberine; Type 2 diabetes; Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Berberine; Metformin

INTERVENTIONS:
Drug: Berberine
Drug: Metformin

SUMMARY:
The purpose of this study is to determine whether berberine is effective in the treatment of type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes is health threats worldwide. However, treatment of this disease is limited by availability of effective medicines. All of the existing oral hypoglycemic agents have secondary failure after long term administration. Thus, new oral medicines are needed for long term control of blood glucose in patients with type 2 diabetes. In diabetes care, dietary approaches have drawn more and more attention in the prevention and treatment of hyperglycemia. Generally regarded as safe (GRAS) plants have been widely used for their benefits in antioxidation, anti-inflammation, anticancer, anti-obesity and anti-diabetes. Numerous botanical products such as pigments that include anthocyanins and flavonoids have been consumed or studied for anti-obesity and anti-diabetes. However, most of these botanical products are mixtures of multiple compounds. It is difficult to control their quality in the study or production. Up to now, as a single purified compound, berberine is demonstrated to have hypoglycemic effect in vitro and in vivo. Berberine is the main active component of Coptis chinensis French, which was used for thousands of years in China in the treatment of human diseases including diabetes.

Comparison(s): Effects of berberine compared with metformin in newly diagnosed type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* HbA1c > 7.0% or FBG > 7.0 mmol/L
* Stable or worsening glycemic control for at least 3 months

Exclusion Criteria:

* Liver damage
* Kidney damage

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-01; Study Completion 2004-12

PRIMARY OUTCOMES:
HbA1c at 13 weeks

SECONDARY OUTCOMES:
Blood glucose at 13 weeks
Blood lipids at 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yin, MD, PhD, Principal Investigator — Department of Endocrinology, Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- Department of Endocrinology, Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China